CLINICAL TRIAL: NCT06008015
Title: An Open-label, Randomized, Fed, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1015" and Co-administration of "BR1015-1" and "BR1015-2" in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1015" and Co-administration of "BR1015-1" and "BR1015-2" Under Fed Conditions in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FIC-CT-102
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR1015 (Experimental)
  Interventions: Drug: BR1015
- BR1015-1 + BR1015-2 (Active Comparator)
  Interventions: Drug: BR1015-1; Drug: BR1015-2

INTERVENTIONS:
Drug: BR1015 — One tablet administered alone
  Arms: BR1015
Drug: BR1015-1 — One tablet administered alone
  Arms: BR1015-1 + BR1015-2
Drug: BR1015-2 — One tablet administered alone
  Arms: BR1015-1 + BR1015-2

SUMMARY:
The purpose of this clinical trial is to evaluate the pharmacokinetics and the safety after administration of "BR1015" and co-administration of "BR1015-1" and "BR1015-2" under fed conditions in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who weigh 50 kg or more and have body mass index (BMI) within the range of 18.0 to 30.0kg/m2 at screening visit.
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial* from the date of the first administration of the investigational products to 14 days after the last administration and disagrees to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken drugs concerned about affecting this clinical trial within 10 days prior to the first day of administration. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs)
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 6 months prior to the first administration date.(However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrointestinal surgery or gastrointestinal diseases that may affect the absorption of drugs. (Except for simple appendectomy, hernia surgery)
* In the case of a female subject, those suspected pregnancy, pregnant woman, lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
AUCτ | 0-72 hours after administration
  Area under the concentration-time curve from time zero to time τ
Cmax | 0-72 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No